CLINICAL TRIAL: NCT01770249
Title: Evaluation of a Novel Endoscopic Treatment for Achalasia: Per-oral Endoscopic Esophagomyotomy (POEM)
Brief Title: Evaluation of a Novel Endoscopic Treatment for Achalasia
Acronym: POEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 03-12-10
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Achalasia
Keywords: dysphagia
MeSH Terms: conditions — Esophageal Achalasia; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- POEM procedure (Other): An endoscopic surgical procedure for achalasia; Per-oral Endoscopic Esophagomyotomy (POEM)will be performed. The POEM procedure will be performed in the operating room under general anesthesia and a scope will then be inserted into your mouth and down your throat and measurements will be taken. With the use of this lighted flexible scope the surgeon will make a small incision in the inner lining of your esophagus (throat), create a tunnel and then cut the muscle between the esophagus (throat) and the stomach. The initial little opening will be closed with a small clip. This procedure will allow easier passage of food into the stomach.
  Interventions: Procedure: Per-oral Endoscopic Esophagomyotomy (POEM)

INTERVENTIONS:
Procedure: Per-oral Endoscopic Esophagomyotomy (POEM) — The surgeon is cutting only through the innermost layers of muscles in the esophagus down to the stomach, leaving the outer layer intact.
  Other Names: POEM

SUMMARY:
This study is to evaluate outcomes of a less invasive surgical procedure for the treatment of achalasia.

DETAILED DESCRIPTION:
This study will assess the feasibility and efficacy of a novel endoscopic procedure, Per-oral Endoscopic Esophagomyotomy (POEM)in treating patients with achalasia.

ELIGIBILITY:
Inclusion Criteria:

* o Subjects with a manometric/radiologic diagnosis of primary achalasia; EGD shows no neoplasm

  * Ability to undergo general anesthesia
  * The subject is > 18 yrs.of age
  * Ability to give informed consent

Exclusion Criteria:

* o Sigmoid achalasia

  * Contraindicated for EGD
  * Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The success of the POEM procedure is measured by improved symptoms as compared to pre-op, including the ability to swallow with low incidence of GERD and significantly reduced resting LES pressure | Within the first 3 months after surgery
  Will assess the outcomes and efficacy of the endoscopic procedure, Per-oral Endoscopic Esophagomyotomy(POEM)in the treatment of achalasia. The patient will be assessed for improvement of their swallowing as assessed on the repeat time barium swallow and increase oral intake without nausea and vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Ponsky Jeffrey, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States